CLINICAL TRIAL: NCT00101192
Title: A Limited Access Phase II Trial of Cetuximab (C225, NSC #714692) in Combination With Cisplatin (NSC #119875) in the Treatment of Advanced, Persistent, or Recurrent Carcinoma of the Cervix
Brief Title: Cetuximab and Cisplatin in Treating Patients With Advanced, Persistent, or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG-0076DD; BMS-CA225-075; CDR0000405839
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical small cell carcinoma; cervical squamous cell carcinoma; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cetuximab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also help cisplatin work better by making tumor cells more sensitive to the drug. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with cisplatin may be a better way to block tumor growth.

PURPOSE: This phase II trial is studying how well giving cetuximab together with cisplatin works in treating patients with advanced, persistent, or recurrent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of cetuximab and cisplatin, in terms of objective tumor response (partial and complete), in patients with advanced, persistent, or recurrent carcinoma of the cervix.
* Determine the nature and degree of toxicity of this regimen in these patients.

Secondary

* Determine the progression-free survival and overall survival of patients treated with this regimen.
* Correlate epidermal growth factor receptor expression with progression-free survival, overall survival, and response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15 and cisplatin IV on days 1 and 8. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 28-62 patients will be accrued for this study within 9-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous or non-squamous cell carcinoma of the cervix

  * Advanced, persistent, or recurrent disease
  * Documented disease progression
* Not amenable to curative therapy
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* At least 1 target lesion

  * Tumors within a previously irradiated field are designated as non-target lesions unless progression is documented or a biopsy is obtained ≥ 90 days after completion of radiotherapy to confirm persistence

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No significant history of cardiac disease within the past 6 months, including the following:

  * Unstable angina
  * Uncontrolled hypertension
  * Uncontrolled congestive heart failure
  * Uncontrolled arrhythmia

Neurologic

* No uncontrolled seizure disorder
* No active neurological disease
* No neuropathy (sensory and motor) > grade 1

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior anti-epidermal growth factor receptor (EGFR) antibody therapy
* No prior chimerized or murine monoclonal antibody therapy

Chemotherapy

* Not specified

Endocrine therapy

* At least 1 week since prior anticancer hormonal therapy
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery

* More than 30 days since prior major surgery, except diagnostic biopsy

Other

* Recovered from all prior therapy
* No prior cytotoxic therapy for cervical cancer
* No prior tyrosine kinase inhibitor therapy that targets the EGFR pathway
* No prior cancer treatment that would contraindicate study therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-09; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Farley, MD, Study Chair — Uniformed Services University of the Health Sciences
Locations (18):
- United States (18):
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Result] Farley J, Sill MW, Birrer M, Walker J, Schilder RJ, Thigpen JT, Coleman RL, Miller BE, Rose PG, Lankes HA. Phase II study of cisplatin plus cetuximab in advanced, recurrent, and previously treated cancers of the cervix and evaluation of epidermal growth factor receptor immunohistochemical expression: a Gynecologic Oncology Group study. Gynecol Oncol. 2011 May 1;121(2):303-8. doi: 10.1016/j.ygyno.2011.01.030. Epub 2011 Feb 16. PMID 21329967

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab: Cetuximab weekly (Cycle 1, day 1 initial loading dose of 400 mg/m2 IV. All subsequent Cetuximab doses are 250 mg/m2 IV) combined with Cisplatin on day 1 and day 8 (30 mg/m2) (one cycle will be three weeks) until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Cetuximab
Started | 76
Completed | 69
Not Completed | 7
Not completed — Ineligible | 6
Not completed — Inevaluable | 1

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.2)
Age, Customized [Number; unit: participants]
  20-29 years | 1
  30-39 years | 11
  40-49 years | 18
  50-59 years | 26
  60-69 years | 9
  70-79 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 69
Cell Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 21
  Clear Cell Carcinoma | 1
  Mucinous Adenocarcinoma | 1
  Adenosquamous | 5
  Squamous Cell Carcinoma | 41

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Per GOG Response Evaluation Criteria In Solid Tumors(RECIST) Criteria:
  Complete Response(CR): disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart.
  Partial Response(PR): at least a 30% decrease in the sum of longest dimensions(LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of nontarget lesions and no new lesions.
  Increasing Disease: at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
  Stable Disease: any condition not meeting the above criteria.
  Indeterminate for response: as having no repeat tumor assessments following initiation of study therapy for reasons unrelated to symptoms or signs of disease.
Time Frame: up to 6 months from study entry
Population: Eligible and evaluable participants
Measure: Number; unit: participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 69
participants
  Complete Response | 1
  Partial Response | 7
  Increasing Disease | 17
  Stable Disease | 34
  Indeterminate | 10

2. Secondary Outcome: Progression-free Survival and Overall Survival at 6 Months After Completion of Treatment
Time Frame: up to 5 years from study entry
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: from study entry up to 5 years
Description: All Adverse Events(AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events(SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 33/69
Other Adverse Events (participants affected / at risk) | 66/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=69)
Death No Ctcae Term - Disease Progression Nos (General disorders) | 2
Fistula, Gi - Ileum (Gastrointestinal disorders) | 1
Obstruction, Gi - Colon (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 2
Hemorrhage/Bleeding - Other (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 2
Opportunisitic Inf Assoc. W/Gr 2 Lymphopenia (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 1
Creatinine (Metabolism and nutrition disorders) | 2
Ggt (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Pain - Other (General disorders) | 1
Pain: Extremity-Limb (General disorders) | 1
Pain: Muscle (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction, Gu - Urethra (Renal and urinary disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 2
Fistula, Gu - Vagina (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 3
Thrombosis/Thrombus/Embolism (Vascular disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=69)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 9
Otitis Middle Ear (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 8
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 13
Platelets (Blood and lymphatic system disorders) | 13
Leukocytes (Blood and lymphatic system disorders) | 23
Hemolysis (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 50
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 4
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 3
S/N Arrhythmia: Atrial Tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 4
Hypotension (Cardiac disorders) | 4
Cardipulmonary Arrest (Cardiac disorders) | 1
Inr (Vascular disorders) | 2
Fibrinogen (Vascular disorders) | 2
Ptt (Vascular disorders) | 3
Sweating (General disorders) | 5
Fever (General disorders) | 10
Weight Loss (General disorders) | 8
Rigors/Chills (General disorders) | 5
Fatigue (General disorders) | 53
Insomnia (General disorders) | 6
Nail Changes (Skin and subcutaneous tissue disorders) | 2
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 14
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 25
Rash (Skin and subcutaneous tissue disorders) | 38
Dry Skin (Skin and subcutaneous tissue disorders) | 11
Decubitus (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7
Burn (Skin and subcutaneous tissue disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1
Hand-Foot (Skin and subcutaneous tissue disorders) | 6
Hot Flashes (Endocrine disorders) | 6
Masculinization Of Female (Endocrine disorders) | 1
Fistula, Gi - Rectum (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 8
Dental: Teeth (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 8
Distention (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 12
Stricture, Gi - Colon (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 29
Anorexia (Gastrointestinal disorders) | 35
Dehydration (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 41
Nausea (Gastrointestinal disorders) | 44
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 20
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 8
Hemorrhage, Gi - Rectum (Vascular disorders) | 6
Hemorrhage, Gu - Ovary (Vascular disorders) | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 5
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 4
Hemorrhage, Gi - Abdomen Nos (Vascular disorders) | 1
Petechiae (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Uterus (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 2
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 2
Inf Unknown Anc: Nose (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 11
Infection - Other (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 1
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 8
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 14
Ast (Metabolism and nutrition disorders) | 6
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 4
Cholesterol,serum High (Metabolism and nutrition disorders) | 2
Proteinuria (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 22
Ggt (Metabolism and nutrition disorders) | 1
Alt (Metabolism and nutrition disorders) | 10
Alkaline Phosphatase (Metabolism and nutrition disorders) | 19
Bilirubin (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 20
Cpk (Metabolism and nutrition disorders) | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 3
Amylase (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 24
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 24
Hypokalemia (Metabolism and nutrition disorders) | 22
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 27
Myositis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Extremity-Upper (Function) (Musculoskeletal and connective tissue disorders) | 1
Gait/Walking (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 5
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 4
Muscle Weakness - Left-Sided (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 5
Pyramidal Tract Dysfunction (Nervous system disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 23
Mood Alteration - Anxiety (Nervous system disorders) | 11
Tremor (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 9
Neuropathy,cranial - Cn Xii Motor-Tongue (Nervous system disorders) | 1
Neuropathy,cranial - Cn Ix Motor-Pharynx (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 25
Neuropathy-Motor (Nervous system disorders) | 1
Dry Eye (Eye disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 1
Blurred Vision (Eye disorders) | 15
Pain - Other (General disorders) | 2
Pain: Pelvis (General disorders) | 6
Pain: Breast (General disorders) | 1
Pain: Vagina (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 2
Pain: Chest Wall (General disorders) | 1
Pain: Throat/Pharynx/Larynx (General disorders) | 3
Pain: Head/Headache (General disorders) | 15
Pain: Neck (General disorders) | 1
Pain: Extremity-Limb (General disorders) | 15
Pain: Buttock (General disorders) | 1
Pain: Back (General disorders) | 20
Pain: Joint (General disorders) | 7
Pain: Bone (General disorders) | 2
Pain: Kidney (General disorders) | 1
Pain: Bladder (General disorders) | 3
Pain: Stomach (General disorders) | 2
Pain: Rectum (General disorders) | 1
Pain: Oral Cavity (General disorders) | 1
Pain: Esophagus (General disorders) | 1
Pain: Dental/Teeth/Peridontal (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 23
Pain: Skin (General disorders) | 1
Pain: Tumor (General disorders) | 2
Pain: Muscle (General disorders) | 4
Pain: Neuralgia (General disorders) | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 2
Airway Obstruction - Bronchus (Respiratory, thoracic and mediastinal disorders) | 1
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 2
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21
Renal/Genitourinary - Other (Renal and urinary disorders) | 2
Leak, Gu - Vagina (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 4
Incontinence, Urinary (Renal and urinary disorders) | 2
Fistula, Gu - Vagina (Renal and urinary disorders) | 1
Fistula, Gu - Bladder (Renal and urinary disorders) | 2
Bladder Spasm (Renal and urinary disorders) | 2
Renal Failure (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 7
Vaginal Discharge (Reproductive system and breast disorders) | 2
Flu-Like Syndrome (General disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 6
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No